CLINICAL TRIAL: NCT00692471
Title: Assessment of Objective Sleep Disturbances in Orthostatic Intolerance Using Actigraphy
Brief Title: Sleep Actigraphy in Postural Tachycardia Syndrome (POTS)
Status: Active, not recruiting | Type: Observational
Sponsor: Satish R. Raj (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Satish R. Raj, Assistant Professor of Medicine & Pharmacology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 080233; K23RR020783 (NIH)
Record Dates: First submitted 2008-06-02; First posted 2008-06-06 (Estimated); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Postural Tachycardia Syndrome; Orthostatic Intolerance; Sleep Disorders
Keywords: Sleep; Orthostatic tachycardia; POTS
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Orthostatic Intolerance; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients meeting the diagnostic criteria for the Postural Tachycardia Syndrome, a form of Orthostatic Intolerance
  Interventions: Device: Actigraphy Watch (motion sensors) with light sensors - ActiWatch from Minimitter
- 2: Healthy control subjects who do not meet the criteria for the Postural Tachycardia Syndrome
  Interventions: Device: Actigraphy Watch (motion sensors) with light sensors - ActiWatch from Minimitter

INTERVENTIONS:
Device: Actigraphy Watch (motion sensors) with light sensors - ActiWatch from Minimitter — Watch to be worn on wrist for 7 days (except in water) that will measure activity/movement.
  Other Names: ActiWatch from Minimitter

SUMMARY:
We propose to use actigraphy (measured by activity watches) as a tool to quantify sleep disturbances in patients with orthostatic intolerance compared with healthy control subjects. In this pilot study, we will test the null hypothesis (Ho) that there are no differences in the sleep quality between patients with orthostatic intolerance and healthy control subjects.

DETAILED DESCRIPTION:
We propose to use actigraphy (measured by activity watches) as a tool to quantify sleep disturbances in patients with orthostatic intolerance compared with healthy control subjects. In this pilot study, we will test the null hypothesis (Ho) that there are no differences in the sleep quality between patients with orthostatic intolerance and healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with orthostatic intolerance by the Vanderbilt Autonomic Dysfunction Center
* Control subjects will be free of orthostatic intolerance and other major medical problems, free of medications during the study
* Age between 18-65 years
* Male and female subjects are eligible.
* Able and willing to provide informed consent

Exclusion Criteria:

* Overt cause for postural tachycardia (such as acute dehydration)
* Self-report of pregnancy
* Inability to give, or withdrawal of, informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with the Postural Tachycardia Syndrome. The criteria include:
  * an increase in heart rate on standing (from supine) of >30 bpm
  * in the setting of symptoms of cerebral hypoperfusion that are worse with standing and better when recumbent
  * the symptoms are daily or almost daily
  * the symptoms are chronic (lasting greater than 6 motnsh)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-06; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Sleep Latency | 1 week

SECONDARY OUTCOMES:
Sleep Efficiency | 1 week
Wake After Sleep Onset | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt Autonomic Dysfunction Center Website — https://www.vumc.org/autonomic-dysfunction-center/vanderbilt-autonomic-dysfunction